CLINICAL TRIAL: NCT05103410
Title: Impact of Preoperative Aripiprazole on Postoperative Analgesia in Laparoscopic Hysterectomy: A Randomized Controlled Clinical Trial
Brief Title: Impact of Aripiprazole on Postoperative Analgesia in Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R 175/2021
Record Dates: First submitted 2021-10-22; First posted 2021-11-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; Analgesia; Hysterotomy
MeSH Terms: conditions — Agnosia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole (Active Comparator): Patients will receive Aripiprazole 30 mg tablet orally 3 h before surgery
  Interventions: Drug: ARIPiprazole 30 MG
- Placebo (Placebo Comparator): Patients will receive placebo tablet which is identical in appearance, size, shape, and color to aripiprazole 3 h before surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARIPiprazole 30 MG — Patients will receive Aripiprazole 30 mg tablet orally 3 h before surgery
  Arms: Aripiprazole
Drug: Placebo — Patients will receive placebo tablet which is identical in appearance, size, shape, and color to aripiprazole 3 h before surgery
  Arms: Placebo

SUMMARY:
The analgesic effect of perioperative use of aripiprazole has not been fully investigated.

So, this study aims to test the effects of aripiprazole versus placebo in reducing postoperative pain following laparoscopic hysterectomy and to explore the potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Physical status American Society of Anesthesiologist (ASA) I or II
* Electively scheduled for laparoscopic hysterectomy,

Exclusion Criteria:

* Patients who refuse to participate
* Body mass index (BMI) > 30
* ASA physical status > II
* Diabetes
* Major illnesses (e.g., cardiac, respiratory, renal, hepatic or neurological)
* Coagulation abnormalities
* Pregnancy
* Known hypersensitivity to aripiprazole or contraindications to its use (a psychiatric illness, patients on antidepressants, dementia-related psychosis)
* History of drug addiction or alcohol abuse
* Mental retardation interfering with the evaluation of pain scores or PCA programs .

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | First 24 hours postoperatively
  After extubation, an intravenous patient-controlled analgesia system, will be connected to the patient (Accufuser Plus® 100 ml, Woo Young Medical Co, Korea) will be prepared with 60 ml normal saline containing 60 mg morphine, it will be programmed to give and 0.5 ml bolus dose with lockout interval of 8 minutes. Time to first Bolus will be estimated considering extubation time is the zero time.

SECONDARY OUTCOMES:
Total opioid consumption | First 24 hours postoperatively
  Total morphine consumption per twenty four hours will be estimated
Visual analogue scale (VAS) | First 24 hours postoperatively
  Pain scores will be evaluated by a blinded observer anesthesiologist at the time of arrival in the PACU, and 10, 20, 30 minutes, 1 h, 2h, 4, 6, 8, 10, 12, 16 and 24 hr thereafter using visual analogue scale (VAS) (0-10 cm: 0 = no pain, 10 = the worst pain possible). The patients will be instructed about usage of VAS preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alansary AM, Elbeialy MAK. Impact of Preoperative Aripiprazole on Postoperative Analgesia in Laparoscopic Hysterectomy: A Randomized Double-blind Placebo-controlled Trial. Clin J Pain. 2024 Jun 1;40(6):341-348. doi: 10.1097/AJP.0000000000001210. PMID 38450551